CLINICAL TRIAL: NCT04548427
Title: Active Controlled, Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-352 Eye Drops in Patients With Dry Eye Disease
Brief Title: Study to Evaluate the Efficacy and Safety of CKD-352
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A100_01DED1924
Record Dates: First submitted 2020-09-10; First posted 2020-09-14 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye Disease; CKD-352
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD-352 (Experimental)
  Interventions: Drug: CKD-352
- Diquafosol Sodium 3% (Active Comparator)
  Interventions: Drug: Diquafosol Sodium 3%

INTERVENTIONS:
Drug: CKD-352 — Eye Drop
  Arms: CKD-352
Drug: Diquafosol Sodium 3% — Eye Drop
  Arms: Diquafosol Sodium 3%

SUMMARY:
The purpose of this study is to compare the efficacy and safety of CKD-352 in patients with dry eye disease

DETAILED DESCRIPTION:
Active controlled, randomized, double-blind, multi-center, phase 3 trial to evaluate the efficacy and safety of CKD-352 eye drops in patients with dry eye disease

ELIGIBILITY:
Inclusion Criteria:

1. More than the age of 19 years old
2. Subjects with dry eye symptoms for at least 3 month
3. Subjects who sign on an informed consent form willingly

Exclusion Criteria:

1. Subjects who have clinically significant ocular surface diseases, abnormal corneal susceptibility and abnormal epiphora
2. Subjects who have clinically significant medical history of ocular disability
3. Subjects who have malignant tumor within 5 years
4. Subjects with known hypersensitivity to investigational product
5. Women who are nursing, pregnant or planning pregnancy during the study
6. Subjects who have received any other investigational product
7. Impossible subjects who participate in clinical trial by investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Changes in Corneal Staining from Baseline and at Week 4 | Baseline, Week 4

SECONDARY OUTCOMES:
Changes in Corneal Staining from Baseline and at Week 2 | Baseline, Week 2
Changes in Conjunctival Staining from Baseline and at Week 2,4 | Baseline, Week 2,4
Changes in Tear Break-up Time from Baseline and at Week 2, 4 | Baseline, Week 2,4
Changes in Schirmer I Test from Baseline and at Week 2, 4 | Baseline, Week 2,4
Changes in Ocular Surface Disease Index from Baseline and at week 2, 4 | Baseline, Week 2,4

CONTACTS AND LOCATIONS:
Overall Officials: Jong Su Lee, M.D, Ph.D, Study Chair — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Pusan, South Korea

IPD SHARING:
Plan to Share IPD: No